CLINICAL TRIAL: NCT01977599
Title: A Randomised Controlled Trial Investigating the Efficacy and Effectiveness of Text Message Reminders to Improve Uptake of Breast Screening by Prevalent Women Living in the London Borough of Hillingdon
Brief Title: Are Text Message Reminders an Effective Intervention for Improving the Uptake of Breast Screening?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 7114/P21R; 12/EM/0418 (Other: NRES Committe East Midlands - Derby)
Record Dates: First submitted 2013-10-09; First posted 2013-11-06 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Breast Screening
Keywords: Text message reminders; Short Message Service (SMS) Reminders; Social Health Inequalities; Breast Screening; Screening; Public Health Intervention; Missed Appointments; Non-attendance

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- No Text Message Reminder (Control) Arm (No Intervention): Control Arm, in which patients are invited to breast screening as per standard West of London Breast Screening Protocol (i.e. without a text message appointment reminder). Uptake of breast screening in this group will be compared with the text message reminder group to test for significant differences.
- Text Message Reminder Arm (Experimental): Patients randomly allocated to this arm of the study will be sent a text message reminding them of the time, date and venue of their breast screening appointment 48 hours in advance.
  Interventions: Other: Text Message Reminder for Breast Screening Appointment

INTERVENTIONS:
Other: Text Message Reminder for Breast Screening Appointment — Non-clinical/administrative.
  Other Names: iPlato Patient Care Messaging will be used to send the text message reminder to the patient.
  Arms: Text Message Reminder Arm

SUMMARY:
Breast Cancer is the single most common cancer, and the third leading cause of cancer cancer deaths, in the United Kingdom. Breast screening is able to detect breast cancer in the early stages of development, during which time it is more easily treatable. Unfortunately, many patients do not attend screening, and surveys issued to these women consistently report "forgetfulness" as the primary reason for missing the appointment. Both telephone reminders and postal reminders have been shown to reduce non-attendance, however, these are time consuming and expensive.

Mobile telephones are becoming an increasingly popular tool for communication between healthcare professionals and patients, one which might offer an inexpensive solution for delivering reminders. Text message reminders have been able to prevent missed appointments in other areas of healthcare, and the same might be true for breast screening.

The investigators are conducting a trial to confirm whether this is the case or not.

In this trial, the investigators will send some women a text message to reminder them of their appointment, and other women no reminder for their appointment. The investigators will then compare the number of women in each group that went to their breast screening appointment.

DETAILED DESCRIPTION:
Breast cancer is the single most common cancer in the United Kingdom, accounting for 16% of all cancer incidences and 7% of all cancer deaths. Fortunately, the natural progression of this malignancy can be beneficially changed through mammographic screening techniques, which enable early detection and treatment of benign and malignant breast disease. However, the success of screening programmes depends not only on the analytical specificity and sensitivity of the screening test itself, but also its ability to attract the "at risk" population. In the United Kingdom, the National Health Service Breast Screening Programme attracts about three quarters of the invited population every three years. In the last screening round (2007-2010), all but one region reported a triennial coverage of more than 75%; London was the exception, reporting a regional coverage of 69%. London consistently fails to meet the national target.

Missed appointments are a primary cause of inefficiency in healthcare delivery, with adverse clinical implications for the non-attending patient, and substantial monetary costs to the health service. To ensure the future success of the breast screening programme it is imperative that strategies for improving uptake of hard to reach populations be developed. Research has demonstrated that receiving an appointment reminder by text message has been successful in improving uptake in other areas of healthcare; the same might be true for breast screening.

Primary Aim: To establish whether text message reminders can significantly improve the uptake of breast screening by women on an "intention-to-treat" basis in the London Borough of Hillingdon.

Secondary Aim: To evaluate whether text message reminders are an effective intervention for improving uptake of the breast screening programme by hard to reach patients such as women living in deprived areas, and those of Black and Minority ethnic backgrounds.

Methodology: A single blind randomised controlled trial evaluating the effectiveness, efficacy, and acceptability of sending a text message appointment reminder to prevalent women (women aged 47-53 years) living in the London Borough of Hillingdon 48 hours prior to their first breast screening appointment. 2,239 women without a history of breast screening, implant, or bilateral mastectomy were included in the study and randomly assigned in a 1:1 ratio to either the control group (n= 1,118) or the intervention group (n= 1,121). Women in the control group were invited to screening but received no reminder for their appointment, whilst women in the intervention group received a text message reminder 48 hours in advance. All women received an information letter about the study with their invitation from the West of London Breast Screening Service, which included a patient "opt-out" request form. Patients were not told whether they would be receiving a text message reminder or not. iPlato Patient Care Messaging was used to deliver the text-message reminders.

ELIGIBILITY:
Inclusion Criteria:

Women aged 47-53 years, being invited for their first breast screen, without a history of breast disease or malignancy, living in the London Borough of Hillingdon, were eligible for inclusion in the trial.

Exclusion Criteria:

Women with a history of breast disease, malignancy, bi-lateral mastectomy, or breast screen, aged over 54 years were not eligible for inclusion in the trial. Non-routine appointments, male appointments, and self referrals were also not eligible for inclusion.

Ages: 47 Years to 53 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2240 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Friedman, FFPH, Study Chair — London Borough of Sutton; Heema Shukla, PhD, Study Chair — Public Health England; Deborah Cunningham, MBBS, Study Chair — Imperial College Healthcare NHS Trust; Robert S Kerrison, BSc, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Charing Cross Hospital, Hammersmith, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Text Message Reminder (Control) Arm | Text Message Reminder Arm
Started | 1118 | 1122
Completed | 1118 | 1122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Text Message Reminder (Control) Arm | Text Message Reminder Arm | Total
Number analyzed (Participants) | 1118 | 1122 | 2240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1118 | 1122 | 2240
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1118 | 1122 | 2240
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1118 | 1122 | 2240

OUTCOME MEASURES:

1. Primary Outcome: Attendance at Breast Screening
Description: Number of women that participate in breast screening in the control (no text message reminder) compared with the number of women that participate in the intervention (text message reminder 48 hours before appointment).
Time Frame: The text message was sent 48 hours before the appointment, attendance was assessed 60 days after the appointment date.
Measure: Count of Participants; unit: Participants
Arm/Group | No Text Message Reminder (Control) Arm | Text Message Reminder Arm
Number analyzed (Participants) | 1118 | 1122
Participants | 661 | 722
Statistical Analysis 1: Comparison: No Text Message Reminder (Control) Arm vs Text Message Reminder Arm; Test type: Other — Chi Square; p < 0.001, Chi-squared

2. Secondary Outcome: Mobile Prevalence
Description: Number of women with a valid mobile telephone number on the GP Clinical System
Time Frame: The accuracy of patient mobile records was assessed for the intervention group at the time the text reminder was sent (i.e. 48 hours before the appointment). A check for the control group was performed at the same time.
Measure: Count of Participants; unit: Participants
Arm/Group | No Text Message Reminder (Control) Arm | Text Message Reminder Arm
Number analyzed (Participants) | 1118 | 1122
Participants | 435 | 456

ADVERSE EVENTS:
Arm/Group | No Text Message Reminder (Control) Arm | Text Message Reminder Arm
All-Cause Mortality (participants affected / at risk) | 0/1118 | 0/1122
Serious Adverse Events (participants affected / at risk) | 0/1118 | 0/1122
Other Adverse Events (participants affected / at risk) | 0/1118 | 0/1122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No